CLINICAL TRIAL: NCT03900156
Title: A Goal-setting With Mentoring Lifestyle Modification Intervention to Reduce Risk of Dementia in Later Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tzu-Ting Huang (Other)
Responsible Party: Sponsor-Investigator, Tzu-Ting Huang, Professor, School of Nursing, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201701926B0
Record Dates: First submitted 2019-03-14; First posted 2019-04-02 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Risk Reduction Behavior; Reduce Risk of Dementia
MeSH Terms: conditions — Risk Reduction Behavior | interventions — Organizational Objectives

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- comparison group (No Intervention): The CG received no extra care.
- Intervention Group (Experimental): Intervention Group, goal-setting with follow-up, will have a structured goalsetting interview using the Bangor Goal-Setting Interview ; once goals are identified and clearly expressed in accordance with SMART principles (specific, measureable, achievable, realistic, and timed)
  Interventions: Other: goal-setting

INTERVENTIONS:
Other: goal-setting — The interviewer will have access to key information from the initial assessment such as details of identified risks. Areas where the participant would like to make changes or improvements will be identified and prioritized, and up to five specific, realistic and achievable goals will be identified.
  Arms: Intervention Group

SUMMARY:
This is a 5-year project. In the 1st year of this study, a pilot randomized controlled trial evaluating the feasibility and acceptability of a goal-setting behavior change intervention aim at reducing modifiable risk factors for preventing cognitive decline. The aim of 2nd to 5th year of this study to investigate whether this multidomain intervention to optimize self-management of cognitive decline risk factors in older individuals, delivered through a mentor- supported interactive internet platform, can reduce the risk of cognitive decline.

DETAILED DESCRIPTION:
Lifestyle factors playing a role in the development of late-life cognitive decline may be modifiable. There is a need for robust evidence about the potential for prevention of cognitive decline through behavior change interventions.

This study involves the development, implementation and initial testing of a behavior change intervention. At the 1st year, a small-scale randomized controlled trial (RCT) will investigate the implementation of a goal-setting intervention aim at promoting behavior change of personal modifiable risks for cognitive decline in the community for >55 years with at least one of the 7 modifiable risk factors for dementia. These older participants in the community (n = 100) will be randomized to either control (had a discussion regarding health and daily activity) or goal-setting with mentoring (the goal-setting interview involving identification of up to five personal goals of personal modifiable risks). All participants will be reassessed after 12 months. The 2nd to the 5th year, is a multisite, prospective, RCT with 36 months intervention. Recruitment of 300 older people (≥55 years) with at least one of the 7 modifiable risk factors for dementia will take place in Northern Taiwan. Participants randomised to the intervention condition will have access to an interactive internet platform, stimulating self-management of dementia risk factors, with remote mentoring by a mentor.

ELIGIBILITY:
Inclusion Criteria:

* in Northern Taiwan
* at least one of the 8 modifiable risk factors for dementia (Hearing loss, Hypertension, Obesity, Smoking, Depression, Physical inactivity, Social isolation, and Diabetes)
* living independently
* in the local community

Exclusion Criteria:

* can't speak chinese

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-04-14 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
cognition | 5 minutes
  Mini-Mental State Examination
cognition | 10 minutes
  Montreal Cognitive Assessment
objective parameters | 2 minutes
  systolic blood pressure
low-density-lipoprotein | 1 minutes
  low-density-lipoprotein
fasting blood sugar | 1 minutes
  fasting blood sugar
body mass index | 1 minutes
  body mass index
waist-hip ratio | 1 minutes
  waist-hip ratio

SECONDARY OUTCOMES:
physical activity scale for the elderly | 5 minutes
  The first page of the questionnaire provides general instructions and shows an example of a completed item. Respondents should be encouraged to answer each item by circling the correct response. All items refer to activities performed in the previous seven days. "Never" and "No" responses should always be marked to indicate any activities the respondent did not perform during that period.
  The leisure activity items require respondents to first report the number of days per week the activity was performed and then the number of hours per day. Space is also provided for respondents to record the types of activities in which they engaged. These reports should be reviewed before computing PASE scores to ensure that specific sports and recreational activities have been recorded in the appropriate categories.
  In this sample scores ranged from 0 to 361. The mean score was 102.9 (standard deviation = 64.1); the median was 90. Mean scores (and standard deviations).
Senior fitness test | 15 minutes
  The Senior Fitness Test was developed as part of the LifeSpan Wellness Program at Fullerton University, by Dr. Roberta Rikli and Dr. Jessie Jones. As such, the test is sometimes known as the Fullerton Functional Test. It is a simple, easy-to-use battery of test items that assess the functional fitness of older adults. The test describes easy to understand and effective tests to measure aerobic fitness, strength and flexibility using minimal and inexpensive equipment.
  The individual fitness test items involve common activities such as getting up from a chair, walking, lifting, bending, and stretching. The tests were developed to be safe and enjoyable for older adults, while still meeting scientific standards for reliability and validity.
Mediterranean Diet Adherence Screener | 5 minutes
  MEDAS. Schröder et al., 2011
Geriatric Depression Scale-15 | 5 minutes
  A short-form GDS that consisted of 15 questions was the primary outcome measure (Sheikh and Yesavage, 1986). Scores of 0-4 are considered normal; 5-8 indicates mild depression; 9-11 indicates moderate depression; and 12-15 indicates severe depression.
  The Chinese version of the GDS-15 demonstrates high reliability (Liao et al., 1995); in this study, the Cronbach's a is .91.
University of California, Los Angeles, Loneliness Scale | 5 minutes
  A 20-item scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. Participants rate each item as either O ("I often feel this way"), S ("I sometimes feel this way"), R ("I rarely feel this way"), N ("I never feel this way").
control, autonomy, self-realization, pleasure-19 | 5 minutes
  Description: The Quality of Life Scale (CASP-19) uses four domains (i.e., control, autonomy, pleasure and self-realization) to assess the quality of life in individuals in early old age.
  Number of items: 19, including 6 items for control, 5 items for autonomy, 4 items for pleasure and 4 items for self-realization.
  Example of statement/item: "I look forward to each day" Response options: 4-point Likert scale ranging from 0, "never" to 3, "often". Total score: Items are summed, yielding a range from 0 to 57 for the total score (domains are usually not used separately). Higher scores indicate higher levels of satisfaction of quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No